CLINICAL TRIAL: NCT04309812
Title: Transcranial Direct Current to Treat Epilepsy at Home
Status: Enrolling by invitation | Phase: Early Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Robert S Fisher, Maslah Saul MD Professor of Neurology, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB# 47711
Record Dates: First submitted 2020-03-09; First posted 2020-03-16 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Epilepsies, Partial
MeSH Terms: conditions — Epilepsies, Partial | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: Randomized to SHORT or LONG dose tDCS as first treatment
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Since the subject sets the stimulation settings for each day of treatment, it is not possible to employ a full placebo with this device. We will inform the subjects that we are uncertain whether short stimulation of 1 minute is less effective than is longer stimulation of 30 minutes, which is a true statement according to our current state of knowledge. We will use a balanced deck of randomized cards setting the initial treatment arm as SHORT in 15 cases and LONG in 15 cases.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Stimulation (Active Comparator): 1 minute duration of stimulation per day for 30 days
  Interventions: Device: transcranial direct current stimulation (tDCS)
- Long Stimulation (Experimental): 30 minutes duration of stimulation per day for 30 days
  Interventions: Device: transcranial direct current stimulation (tDCS)

INTERVENTIONS:
Device: transcranial direct current stimulation (tDCS) — Electrical stimulation of scalp over a seizure focus

SUMMARY:
This is a placebo-controlled study of the effectiveness of transcranial direct current stimulation (tDCS) at home to reduce seizures and EEG spikes.

DETAILED DESCRIPTION:
Electrical stimulation is a promising new therapy to reduce seizures, but current methods require inserting wires under the skull or into brain. This project will use direct-current electrical stimulation pulses delivered from scalp electrodes to provide stimulation. The goal is to reduce seizures without the need for surgery.

2. PROCEDURES:

2.1. Baseline: Upon signing of consent, subjects will have an initial screening clinic visit with a neurological history and examination. You will record a seizure diary for one month prior to start of stimulation.

2.2. Baseline EEGs: A 2-hour recording will be done with the 256 channel hydrogel electrocap (currently used for clinical studies). Subjects will be maintained awake for consistency, since sleep affects EEG activity.

2.3. Seizure Diary: The subject (and/or family) will maintain a seizure diary during the baseline, treatment, and for one month after their final stimulation treatment. The seizure diary will be reviewed by the study coordinator in a phone contact once per week.

2.4. Baseline antiepileptic drug levels for patients taking phenytoin, phenobarbital, carbamazepine, valproic acid, lamotrigine or levetiracetam.

2.5. Baseline neuropsychological testing: Subjects will take baseline neuropsychological tests, consisting of Beck Depression Index, the National Hospital Seizure Severity Scale, the Personal Impact of Epilepsy (PIES) scale and the Montreal Cognitive Assessment basic scale.

3. Transcranial Direct Current Stimulation Treatment Procedures

3.1. tDCS: The direct current stimulus will be delivered via a commercially-available ActivaDose transcranial direct current stimulator (or if it becomes unavailable, a commercially available Soterix Medical device) through a saline-moistened pad placed over the region of the seizure focus. Cathodal (negative) DC current will be delivered to the seizure focus and anodal (positive) current over the oppositel forehead.

3.2. Ensuring comfort: Direct current stimulation will be at an intensity of 2 mA for 30 minutes per session, with slow ramp-up and ramp down of the current. This level of stimulation is usually comfortable to most subjects. If the sensation is significantly uncomfortable, the stimulation will be reduced to 1 mA, and if that is uncomfortable, you will be discontinued from the study.

3.3. Except for initial, mid-study and final EEG recording and the device use training session, this study will take place in your home. During a training session for home use you will be made familiar with the ActivaDose operation by study staff. Features to be learned will include:

a. Turning on the device b. Setting the stimulation to 2 mA c. Setting the stimulation duration to 1 minute or 30 minutes. Attachment of the 2 pads (cathode and anode). e. Proper placement of pads, careful explanation of cathode to go over the seizure zone.

f. Pad removal, disposal and device storage g. Schedule for treatments

3.4. Placebo: It is not yet clear whether short stimulation of 1 minute (SHORT) is less effective than is longer stimulation of 30 minutes (LONG). A balanced deck of randomized cards setting the initial treatment arm as SHORT in 15 cases and LONG in 15 cases. However, you will receive both treatments in different months, and afterwards will have the option of continuing with the one that works best for you (assuming that one of the treatments helps).

3.5. Schedule: After signing consent, the study will begin with one month of baseline while keeping a daily seizure diary. During this baseline month, you will have baseline EEG recorded and training on device use. There will then be one month of treatment SHORT or LONG, one month no treatment "wash-out," then one-month of treatment LONG or SHORT, including the treatment not given in the first round. Diary will be kept for one month after the second treatment. You will be given a printed schedule of dates and the device settings to use for each date.

3.6. Medications: During the baseline, treatment months, washout month and one month of follow-up after treatment, efforts will be made to keep your seizure medicines constant. However, medicines can be changed if the treating physician believes it is necessary for your welfare

3.7 Visits: Phone visits will be made and logged one week (± 3 days) after initiating treatment SHORT or treatment LONG. Three in-person visits will be performed: at baseline and after completion of the two treatment months.

3.8. Follow-up testing: A 1-hour EEG will be performed during the wash-out month and after completion of both treatment arms. The final EEG will record 2 hours of spontaneous activity, followed by 30 minutes of Active tDCS at 2 mA, and then 30 min of subsequent recording. This will be done to evaluate any acute EEG changes produced by tDCS. Together with the baseline study, this will total 3 EEGs. Neuropsychological tests will be administered twice: at baseline and after completion of all treatments.

3.9. Escape Criteria: For individual subjects, the study will be terminated for any of the following reasons:

1. Unacceptable discomfort or pain in response to the tDCS treatment.
2. A tonic-clonic seizure occurring during a stimulation session.
3. Emergence of a first-in-life tonic-clonic seizure at any time during the study.
4. Generalized status epilepticus.
5. Tripling or more of the baseline seizure frequency.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-100, inclusive.
* Has a clinical diagnosis of epilepsy
* Has at least 4 countable seizures per month
* Has not had control with at least 2 anti-seizure medicines
* Able to maintain a constant medication for duration of the study (rescue meds allowed)
* Subject or legally authorized representative is able to understand consent and keep a seizure diary in English

Exclusion Criteria:

* A disease likely to progress over course of the study
* Psychogenic non-epileptic seizures
* Suicide attempt or psychiatric hospitalization past 2 years
* A skin condition interfering with scalp electrodes or allergy to silver
* Women will verify not pregnant, and if applicable, have a serum pregnancy test

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in seizures per month | Within 1 week of end of the SHORT treatment and within 1 week of end of the LONG treatment
  Number of seizures recorded in the patient diary
Change in seizures per month | Recorded at time of study entry (BASELINE) and within 1 week of end of the SHORT treatment
  Number of seizures recorded in the patient diary
Change in seizures per month | Recorded at time of study entry (BASELINE) and within 1 week of end of the LONG treatment
  Number of seizures recorded in the patient diary

SECONDARY OUTCOMES:
Change in severity of seizures | Within 1 week of end of the SHORT treatment and within 1 week of end of the LONG treatment
  Severity of seizures recorded in the patient diary
Change in duration of seizures | Within 1 week of end of the SHORT treatment and within 1 week of end of the LONG treatment
  Duration of seizures as recorded in the patient diary
Number of epileptiform EEG spikes | Within 1 week of end of the SHORT treatment and within 1 week of end of the LONG treatment
  Count by blinded evaluator on EEGs before and after tDCS

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Stanford Hospital, Stanford, California
  - Stanford University School of Medicine, Stanford, California

IPD SHARING:
Plan to Share IPD: No